CLINICAL TRIAL: NCT04267939
Title: An Open-label Phase 1b Study to Determine the Maximum Tolerated and/or Recommended Phase 2 Dose of the ATR Inhibitor Elimusertib (BAY 1895344) in Combination With PARP Inhibitor Niraparib, in Participants With Recurrent Advanced Solid Tumors and Ovarian Cancer
Brief Title: ATR Inhibitor Elimusertib (BAY1895344) Plus Niraparib Phase 1b Study in Advanced Solid Tumors and Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: There was no anticipated benefit of the experimental combination as tested over available standard therapies; therefore Sponsor has decided to terminate the investigation.
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 18595; 2018-003930-34 (EudraCT Number)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumors (Excluding Prostate Cancer); Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — BAY 1895344; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose escalation of elimusertib_Part A.1 (Experimental): Dose escalation will initiate with Part A.1 in which niraparib is used at a lower fixed dose.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Niraparib
- Dose escalation of elimusertib_Part A.2 (Experimental): If the starting dose level in Part A.1 is tolerated, dose escalation in Part A.2 may be initiated on an optional basis. In Part A.2, niraparib is used at a higher fixed dose.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Niraparib
- Dose expansion_sub-population 1_lower dose of niraparib (Experimental): MTDs and/or candidate RP2Ds for elimusertib used in combination with niraparib at a lower fixed dose.
  MTD: Maximum tolerated dose. RP2D: Recommended phase 2 dose.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Niraparib
- Dose expansion_sub-population 2_lower dose of niraparib (Experimental): MTDs and/or candidate RP2Ds for elimusertib used in combination with niraparib at a lower fixed dose.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Niraparib
- Dose expansion_sub-population 1_higher dose of niraparib (Experimental): MTDs and/or candidate RP2Ds for elimusertib used in combination with niraparib at a higher fixed dose.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Niraparib
- Dose expansion_sub-population 2_higher dose of niraparib (Experimental): MTDs and/or candidate RP2Ds for elimusertib used in combination with niraparib at a higher fixed dose.
  Interventions: Drug: Elimusertib (BAY1895344); Drug: Niraparib

INTERVENTIONS:
Drug: Elimusertib (BAY1895344) — Elimusertib will be administered in 28-day cycles.
Drug: Niraparib — Niraparib will be administered in 28-day cycles.

SUMMARY:
The purpose of the study is to test how well patients with advanced solid tumors and ovarian cancer respond to treatment with elimusertib in combination with niraparib. In addition researchers want to find for patients the optimal dose of elimusertib in combination with niraparib, how the drug is tolerated and the way the body absorbs, distributes and discharges the drug. The study medication elimusertib works by blocking a substance produced by the body (ATR Kinase) which is important for the growth of tumor cells. Niraparib works by blocking a substance produced by the body (PARP enzymes) in a way that tumor cells can be killed, or made more susceptible to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age, at the time of signing the informed consent.
* Participants must have histologically confirmed diagnosis of the following indications as described below:

  * Dose escalation (Part A): recurrent advanced solid tumors, excluding prostate cancer, who experienced disease progression after treatment with standard of care therapy for metastatic disease.
  * Dose expansion (Part B): recurrent EOC, fallopian tube or primary peritoneal cancer

    * Sub-population 1: participants PARPi naïve and with a platinum-resistant/refractory disease (recurrence with a PFI < 6 months from last platinum-based regimen). Participants may not have had more than 3 prior therapies since the development of platinum resistance.
    * Sub-population 2: participants with disease progression on PARPi (including niraparib), administered as maintenance as well active line of therapy. Participants must have not received further line of therapy after disease progression on PARPi.
* Participants in dose escalation (Part A) of the study will need to have tumor-associated DDR deficiency and/or CCNE1 gene amplification.

  -- A homozygous deletion and/or a deleterious mutation in a gene reported to be involved in DNA repair and/or sensitive to ATRi's and/or PARPi's.
* Participants in dose expansion (Part B) of the study will need to have tumor associated DDR deficiency (Sub-population 1). Participants in Part B (Sub-population 2) are not enrolled based on the presence or absence of a particular biomarker.
* Participants must have disease progression and measurable disease, as defined by RECIST 1.1.
* Available archival tumor tissue ≤ 12 months old, otherwise a fresh baseline tumor biopsy should be obtained.
* ECOG PS of 0 to 1
* Life expectancy of at least 12 weeks
* Adequate bone marrow function as assessed by the following laboratory tests to be conducted within 7 (±2) days before the first dose of study intervention:

  * Hemoglobin (Hb) ≥ 10 g/dL
  * Platelet count ≥ 150 x 10^9/L
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
* Participants must have adequate organ function.
* Participants must have adequate coagulation.
* Adequate cardiac function per institutional normal measured by echocardiography (recommended) or cardiac MRI per institutional guidelines.
* A female participant is eligible to participate if she is not pregnant (confirmed by a negative serum pregnancy test within 7 (±2) days of first study intervention), not breastfeeding, or is not a woman of childbearing potential (WOCBP). WOCBP must agree to use highly effective contraception during the intervention period and for at least 6 months (180 days) after the last dose of study intervention.

Exclusion Criteria:

* Inability to swallow oral medication
* Known hypersensitivity to elimusertib and/or niraparib or excipients of the preparations or any agent given in association with this study
* History of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) diagnosis
* Ongoing or active uncontrolled infection (bacterial, fungal, or viral; e.g. hepatitis viral) of CTCAE grade ≥ 2 that requires systemic treatment
* Participants with HIV may be be ineligible depending on various parameters, but are not automatically excluded.
* Immunocompromised participants (e.g. diagnosis of immunodeficiency or ongoing immunosuppressive therapy)
* Pleural effusion or ascites that causes respiratory compromise (CTCAE grade ≥ 2 dyspnea)
* Active HBV or HCV infection that requires treatment.
* Moderate or severe hepatic impairment, i.e. Child Pugh Class B or C
* Participants with significant cardiovascular disease and/or relevant findings meeting the below criteria are excluded:

  * History of cardiac disease: congestive heart failure NYHA class > II, unstable angina (angina symptoms at rest), new-onset angina (within the past 6 months before study entry), myocardial infarction within the past 6 months before study entry, or cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers, calcium channel blockers, and digoxin are permitted).
  * Clinically relevant findings in the ECG such as a second- or third-degree atrioventricular block, prolongation of the QRS complex ≥ 120 ms, or prolongation of the of the QTc interval (Fridericia) over 450 ms unless agreed otherwise between the investigator and the sponsor's medically responsible person. QTc > 450 ms detected in 2 or more time points within a 24-hour period are excluded.
  * Clinically significant arterial hypertension despite optimal medical management (per investigator´s opinion). Clinically significant hypertension defined as systolic blood pressure above 150 mmHg and/or diastolic blood pressure above 90 mmHg, despite optimal medical management. For participants taking antihypertensive medication, blood pressure should be stable/ controlled for more than 7 days before first dose of study medication.
* Previous treatment with an ATR Inhibitor
* Participants in Part A and Part B (Sub-population 2): Previous treatment with known or putative PARPi, if discontinued for CTCAE grade ≥ 3 AEs or CTCAE grade ≥ 3 hypersensitivity to PARPi. Participants in Part B Sub-population 1 must not have received prior PARPi treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | Up to 30 days after the last administration of study intervention
Severity of treatment emergent adverse events (TEAEs) | Up to 30 days after the last administration of study intervention
Incidence of treatment emergent serious adverse events (TESAEs) | Up to 30 days after the last administration of study intervention
Severity of treatment emergent serious adverse events (TESAEs) | Up to 30 days after the last administration of study intervention
Maximum tolerated dose (MTD): Frequency of Dose Limiting Toxicities (DLTs) at each dose level during the DLT observation period for Cycle 1 | Cycle 1, 28 days after first administration of study intervention
Recommended Phase II dose (RP2D) of elimusertib | Up to 30 days after last administration of study Intervention

SECONDARY OUTCOMES:
Incidence of participants with complete response (CR) | At baseline and at the start of every 2nd cycle (each cycle is 28 days) starting with Cycle 3, and at the start of every 4th cycle after Cycle 11 up to 24 months.
Incidence of participants with partial response (PR) | At baseline and at the start of every 2nd cycle (each cycle is 28 days) starting with Cycle 3, and at the start of every 4th cycle after Cycle 11 up to 24 months.
Incidence of participants with stable disease (SD) | At baseline and at the start of every 2nd cycle (each cycle is 28 days) starting with Cycle 3, and at the start of every 4th cycle after Cycle 11 up to 24 months.
Incidence of participants with progressive disease (PD) | At baseline and at the start of every 2nd cycle (each cycle is 28 days) starting with Cycle 3, and at the start of every 4th cycle after Cycle 11 up to 24 months.
Objective response rate (ORR) | At baseline and at the start of every 2nd cycle (each cycle is 28 days) starting with Cycle 3, and at the start of every 4th cycle after Cycle 11 up to 24 months.
Disease control rate (DCR) | At baseline and at the start of every 2nd cycle (each cycle is 28 days) starting with Cycle 3, and at the start of every 4th cycle after Cycle 11 up to 24 months.
Cmax (Maximal plasma exposure) of elimusertib after single dose administration | Cycle 1 Day 5 and Cycle 1 Day 21, each cycle is 28 days.
AUC(0-8) of elimusertib after single dose administration | Cycle 1 Day 5 and Cycle 1 Day 21, each cycle is 28 days.
Cmax,md of elimusertib after multiple dose administration | Cycle 1 Day 5 and Cycle 1 Day 21, each cycle is 28 days.
AUC(0-8)md of elimusertib after multiple dose administration | Cycle 1 Day 5 and Cycle 1 Day 21, each cycle is 28 days.
  AUC: Area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Smith G, Alholm Z, Coleman RL, Monk BJ. DNA Damage Repair Inhibitors-Combination Therapies. Cancer J. 2021 Nov-Dec 01;27(6):501-505. doi: 10.1097/PPO.0000000000000561. PMID 34904813